CLINICAL TRIAL: NCT00456248
Title: Phase 4 Study Using Infergen and Ribavirin in Patients With Chronic Hepatitis C Virus Who Achieved Partial Response to Peginterferon-alfa and Ribavirin Therapy
Brief Title: Infergen and Ribavirin Treatment of Patients With HCV Who Achieved Partial Response to Peginterferon-alfa and Ribavirin
Acronym: ENHANCE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VRX-CIFN-402
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis C
Keywords: Chronic Hepatitis C; Liver; Pegylated; Interferon; Ribavirin; Combination; Nonresponder; Relapser; HCV; Infergen; SVR
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — interferon alfacon-1; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Infergen 15 ug QD plus RBV for 36 weeks
  Interventions: Drug: Infergen and ribavirin
- 2 (Experimental): Infergen 15 ug QD plus RBV for 48 weeks
  Interventions: Drug: Infergen and ribavirin
- 3 (Active Comparator)
  Interventions: Drug: Infergen and ribavirin

INTERVENTIONS:
Drug: Infergen and ribavirin — Infergen 15 ug QD plus RBV for 36 weeks and Infergen 15 ug QD plus RBV for 48 weeks

SUMMARY:
This is a 60-to-72 week multicenter study to evaluate Infergen and Ribavirin in patients with Chronic Hepatitis C Virus after partial response to treatment using peginterferon-alfa and Ribavirin therapy. The study will be conducted at approximately 50 sites across the United States.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age and no older than 65 years with compensated chronic HCV infection based on a history of positive serum anti-HCV antibody and/or HCV RNA
* Diagnosed with HCV Genotype 1, 4, 5 or 6 as determined during the screening visit
* The starting doses in the initial treatment must have been 1.5 μg/kg/week PEG-Intron or 180 μg/week Pegasys, and 1000/1200 mg/day ribavirin based on body weight. Patients must have been at least 80% compliant during the initial peginterferon/ribavirin therapy, per patient account.
* Liver biopsy indicating F0-F4 must be performed within 3 years prior to screening. Documentation of the results of the biopsy must be available. If documentation is not available, a liver biopsy must be performed during the screening period. (A maximum of 10 patients in each of the three treatment groups will be patients with a fibrosis score of F4)
* Documented partial response after 12 weeks of treatment as a therapy-naive patient with one course of peginterferon alfa-2a (PEGASYS) and Ribavirin or peginterferon alfa-2b (Peg-INTRON) and Ribavirin

Exclusion Criteria:

* Detectable HCV RNA after 12 weeks if initial peginterferon alfa/ribavirin therapy and <2 log decrease in HCV RNA at Week 12 from baseline.
* HCV Genotype 2 or 3
* Severe neuropsychiatric disorder.
* History or clinical manifestations of significant metabolic, hematological, pulmonary, ischemic heart disease, significant or unstable heart disease, gastrointestinal, neurological, renal, urological, endocrine, ophthalmologic disorders including severe retinopathy, or immune-mediated disease.
* Known HIV infection or positive HIV at screening.
* Pregnant or breast-feeding patients.
* Underlying autoimmune disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the proportion of patients with a sustained viral response (SVR) defined as undetectable serum HCV RNA at the end of the 24 week post-treatment follow-up period. | 1.5 years

SECONDARY OUTCOMES:
Compare proportion of patients with SVR after switching treatment with Infergen/Ribavirin for 48 weeks versus those treated for 36 weeks | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell L Schiffman, MD, Principal Investigator — Virginia Commonwealth University
Locations (4):
- United States (4):
  - Atlantic Gastroenterology Associates, Atlanta, Georgia
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Caroline Digestive Health Associates, Harrisburg, North Carolina
  - Liver Institute at Methodist Dallas, Dallas, Texas